CLINICAL TRIAL: NCT02318576
Title: Computerized Cognition Testing and Cognitive Motor Interference in MS
Acronym: C3PO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Jacob Sosnoff, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 15333
Record Dates: First submitted 2014-12-09; First posted 2014-12-17 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): This group will do nothing for the 12 week program.
- Cognitive Trained Group (Experimental): This group will train three time a week for one hour on the given computerized cognitive training website for the 12 week program.
  Interventions: Other: Cognitive Training

INTERVENTIONS:
Other: Cognitive Training — Computerized Cognitive Training: The online computer training program will be administered on the participants' home computer. The training program will consist of a total of 36 sessions (3 times/week for 12 weeks). Each session will last no more than 60 minutes and consist of five different cognitive exercises designed to improve cognitive processing speed, memory and executive function. All exercises will involve visual stimuli and a motor response (key or button press). Exercises will be adaptive to participants' individual ability and start with minimal difficulty.
  Arms: Cognitive Trained Group

SUMMARY:
This study seeks to examine whether 12 weeks of home-based computerized cognitive training on Cognitive Motor Interference (CMI) will improve walking and cognitive function in persons with MS.

DETAILED DESCRIPTION:
Walking and cognitive impairments are common in persons with multiple sclerosis (MS). Approximately 85% of persons with MS report walking as a major limitation, whereas 65% experience cognitive dysfunction. Traditionally, walking and cognition have been viewed as unrelated, but there is evidence of cognitive-motor interference (CMI). CMI is believed to stem from damage to common neural substances responsible for cognitive and motor functions. Recent evidence supports cognitive-motor interference in persons with MS. For example, there is evidence that walking performance declines when performed in conjunction with a simultaneous cognitive task (i.e., dual task cost [DTC] of walking). This decline in walking performance is greater in persons with MS compared to healthy control and is associated with walking impairment. The degree of CMI during walking is associated with walking performance and cognitive function in people with MS. For instance, CMI has been found to be related to general cognitive function and self-reported everyday cognitive errors in people with MS with minimal disability.

Cognitive-motor interference during mobility tasks is of practical and clinical importance because it has been linked to decreased community mobility and a greater risk of falls in other clinical populations such as stoke, Parkinson's disease and the elderly. We have recently demonstrated that the degree of CMI during walking was associated with physiological fall risk in MS, whereas gait velocity in and of itself was not.

Evidence gathered from other special populations suggests that CMI can be minimized with interventions. However, there is no research on rehabilitation strategies on CMI in people with MS. One possible approach for improving cognitive function and reducing CMI involves computerized cognitive testing. This approach capitalizes on neural plasticity and has been found to improve cognitive function, walking and balance in healthy older adults. Although there is limited preliminary data suggesting this type of training may improve cognitive function in people with MS, there is no extant data indicating computerized cognitive training will impact mobility. Based on association between cognitive and motor function in people with MS, it is possible that cognitive training may lead to improvements in walking performance as seen in other clinical populations. One major advantage of computerized cognitive training is that it can be completed without direct supervision and in one's home to minimize various barriers to clinic-based rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* medically confirmed MS diagnosis, relapse free in the last 30 days, willingness to complete 12 week intervention, a computer with Internet access and capacity to run the cognitive training software, and a willingness to travel twice to our research lab.

Exclusion Criteria:

* Non-ambulatory, inability to see/read computer screen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Cognitive motor interference meausred by the percent change in walking velocity from single (walking only) to dual task (walking while thinking). | 12 weeks
  CMI will be operationalized as the percent change in walking velocity from single (walking only) to dual task (walking while thinking). Participants will complete a total of 4 walking trials over a 20' pressure sensitive (Zeno™) walkway at a comfortable pace. Half of the trials will be conducted while reciting every other letter of the alphabet (i.e. N, P, R, etc). Each trial will start with a different letter to minimize practice effects. The order of the dual task conditions will be counter balanced. Prior to walking trails participants will complete the alternating letter task for two 10-second trials while seated.

SECONDARY OUTCOMES:
Cognitive Function | 12 weeks
  Cognition will indexed at each assessment utilizing the brief international cognitive assessment for MS (BICAMS) which is composed of the symbol digit modalities test (SDMT), California verbal learning test-II (CVLT-II) and the revised brief visuospatial memory test (BVMT). Respectively, these validated tests quantify cognitive processing speed, memory and executive function. All cognitive tests will be performed in an environment free of distractions. We note that these tests are valid and reliable in persons with MS.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob J Sosnoff, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Motor control research lab, Urbana, Illinois, United States